CLINICAL TRIAL: NCT01089465
Title: Cimex Lectularius or Bed Bugs : Vector of Infectious Agents and Pathogenic Role
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 09-API-01
Record Dates: First submitted 2010-03-12; First posted 2010-03-18 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Sting
Keywords: Bed bugs; Cimex; insects; bites
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Collection of the bedbugs and dermatological follow-up of the stings — Collection of the bedbugs and dermatological follow-up of the stings at J1 J7 J14 J21 J28

SUMMARY:
During the last years, the investigators were the witness to the increase of a old emerging pest due to bed bugs (Cimex lectularius) in the world. Insecticides resistances apparitions and internationals transports increases seem to be the reasons of the pest. Cimex lectularius as vector of parasites, bacteria or virus was often suggested although not much observation are recently investigated in France. This study intends to examine the vectorial ability and the direct pathogenicity of Cimex lectularius.

ELIGIBILITY:
Inclusion Criteria:

* On the site of takings presence of insects and eggs evoking bedbugs of beds. The identification of certainty will be made in the laboratory. All the insects not apartment to the family of Cimicidae (Criterion of exclusion) are thrown(cast) in trash cans of laboratories for organic products.
* voluntary Patients after reading of the information sheet and the signature of the consent
* Membership of the patient in the national insurance scheme

Exclusion Criteria

* On the site of takings absence of insects and eggs evoking bedbugs of beds
* During the identification of certainty in the laboratory, the captured insects do not make parties of the family of Cimicidae
* The subjects deprived of freedom.
* Patients cancelling their consent.
* Patients violating the protocol of search(research)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2010-03 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Morphological identification of every bedbug Porterage of bacterial agents Porterage of viral agents Biomolecular identification of the insect A breeding of bedbugs Tests of sensibility in insecticides | day 1

SECONDARY OUTCOMES:
Study of the direct pathogenicity of lectularius C. | day 1, 7, 15 and 30
  During each of four consultations a questionnaire and a descriptive index card(form) of the general and dermatological signs will be informed. The criteria of evaluation, associated with anonimisées photos, are split into two groups: general Signs and dermatological Signs

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Delaunay, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Collection of the bedbugs and dermatological follow-up of the stings, Nice, France